CLINICAL TRIAL: NCT01035073
Title: Functional Change and Efficacy of Duloxetine in Patients With Major Depression and Co-Morbid Soft Tissue Discomfort Symptoms
Brief Title: Functional Change and Efficacy of Duloxetine in Patients With Co-Morbid Depression & Soft Tissue Discomfort Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F1J-US-X018
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Results first posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Major Depressive Disorder; Soft Tissue Discomfort Syndrome; Pain
MeSH Terms: conditions — Depressive Disorder, Major; Pain | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Duloxetine (Experimental)
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — 30-60 mg daily for 8 weeks
  Other Names: Cymbalta

SUMMARY:
The objective of this study is to determine the time course of duloxetine efficacy on the symptoms of Major Depressive Disorder (MDD)and on the symptoms of Soft Tissue Discomfort Syndrome(STDS) via use of 24-hour Actigraph™ measures.

We hypothesize that there will be a reduction in both MDD and STDS symptoms in MDD patients with co-morbid STDS symptoms. We further hypothesize that there will be a rapid improvement in functional outcome ratings and 24-hour activity in MDD patients with co-morbid STDS symptoms which may occur even before the antidepressant effect is observed.

ELIGIBILITY:
Inclusion Criteria:

* > 17 years old
* All races and ethnicity
* DSM IV-TR Axis I diagnosis of MDD
* Co-morbid STDS
* Baseline 17-item Hamilton Depression Rating > 13

Exclusion Criteria:

* Primary Axis I disorder other than MDD
* History of mania or psychosis
* Actively suicidal
* Required hospitalization
* A alcohol or substance abuse or dependence within the preceding 3 months
* Pregnant or nursing
* Unstable medical condition (other than STDS)
* Narrow-angle glaucoma
* Sensitivity to duloxetine, concurrent antidepressant, tranquilizer, or mood stabilizer use
* Hepatic or renal insufficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay D Amsterdam, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Depression Research Unit, University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Depression Research Unit — http://www.med.upenn.edu/dru

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The investigator has succumb to serious health issues which prevents him from physically inputting data in the system. The study team is no longer at the university and despite all efforts to contact them in order to enter data on the investigator's behalf, data are not available.
Period: Overall Study
Arm/Group | Duloxetine
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The investigator has succumb to serious health issues which prevents him from physically inputting data in the system. The study team is no longer at the university and despite all efforts to contact them in order to enter data on the investigator's behalf, data are not available.
Arm/Group | Duloxetine
Number analyzed (Participants) | 0
Age, Customized [unit: participants]
Sex/Gender, Customized [unit: participants]
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: 24-hour Activity Level
Time Frame: Baseline and Week One of Treatment
Population: as for baseline characteristics
Arm/Group | Duloxetine
Number analyzed (Participants) | 0

2. Secondary Outcome: Functional Symptom Questionnaire
Time Frame: Baseline; Week 6 and Week 8 of Treatment
Population: as for baseline characteristics
Arm/Group | Duloxetine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 Years
Description: The investigator has succumb to serious health issues which prevents him from physically inputting data in the system. The study team is no longer at the university and despite all efforts to contact them in order to enter data on the investigator's behalf, data are not available.
Arm/Group | Duloxetine
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Data is unavailable for the following reasons:

investigator has succumb to serious health conditions preventing him from entering data, and study team members no longer work for the university and cannot be reached to input data despite efforts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes